CLINICAL TRIAL: NCT03069781
Title: The Effects of 17β-estradiol on Skeletal Muscle Mass Following Immobilization
Brief Title: The Effects of 17β-estradiol on Skeletal Muscle
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, Stuart Phillips, Professor, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: REB-2919
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Muscle Atrophy
Keywords: estrogen
MeSH Terms: conditions — Muscular Atrophy | interventions — Estradiol; Glucans

STUDY DESIGN:
Intervention Model Description: Parallel-group, double-blinded, randomized controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both forms of supplementation (estrogen and placebo) will be packaged and administered in identical fashion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 17β-estradiol (Experimental): 1mg/day for 3-days and 3mg/day for 7-days of 17β-estradiol (Estrace, Acerus Pharmaceuticals Corporation, Mississauga, ON, Canada). 7 Day Breg Knee Brace unilateral immobilization.
  Interventions: Drug: 17β-estradiol
- Placebo (Placebo Comparator): 400 mg/day for 10-days of Polycose (Abbott Laboratories, St. Laurent, QC, Canada).7 Day Breg Knee Brace unilateral immobilization.
  Interventions: Drug: Polycose

INTERVENTIONS:
Drug: 17β-estradiol — 1mg/day for 3-days and 3mg/day for 7-days of Estrance
  Other Names: Estrance
  Arms: 17β-estradiol
Drug: Polycose — 400 mg/day for 10-days of Polycose (Abbott Laboratories, St. Laurent, QC, Canada)
  Other Names: Enteral Nutrition Formulas
  Arms: Placebo

SUMMARY:
The maintenance of skeletal muscle mass and function is critical for healthy aging. Muscle loss with disuse, termed muscle disuse muscle atrophy, leads to impaired functional capacity, the onset of insulin resistance, as well as a heightened risk for morbidity and mortality. With advancing age there is a chronic wasting of muscle. This is especially true in women, where rapid rates of decline in muscle mass and greater anabolic resistance are experienced around the time of menopause, despite higher protein synthesis rates. As women have a longer life expectancy, they are particularly venerable to age-related frailty and morbidity.

Skeletal muscle protein turnover serves to maintain the optimal function of proteins and also provides plasticity of the tissue during altered demands such as during increased loading or unloading of the muscle. Reduced periods of physical activity also have a similar, albeit milder, impact on skeletal muscle and most, people will likely experience multiple bouts of skeletal muscle disuse during their lifetime from which some, particularly older adult women, will fail to fully recover. Thus, muscle disuse atrophy is a significant and continuing problem as reclamation of lost muscle mass, strength/function, and potentially metabolic health (particularly insulin-induced glucose disposal), following disuse is oftentimes incomplete and may be further exacerbated after menopause.

Previous evidence has demonstrated that in the loss of muscle mass is less pronounced in post-menopausal women when receiving hormone replacement therapy. Skeletal muscle has estrogen-β-receptors on the cell membrane, in the cytoplasm and on the nuclear membrane, and therefore a direct mechanistic link between low estrogen levels and a decrease MPS. Interestingly, despite higher rates of protein synthesis, older women still lose muscle mass with advancing age. It has been suggested that the negative muscle protein balance is due to an enhanced rate of MPB. Insulin is a potent inhibitor of MPB and estrogen has been shown to enhance insulin sensitivity in skeletal muscle. However, to our knowledge, no study has examined the efficacy of estrogen supplementation to attenuate the losses of skeletal muscle mass and function during a period of disuse. The findings of this investigation may yield critical data for those who wish to combat skeletal muscle disuse atrophy, particularly after menopause.

DETAILED DESCRIPTION:
Design and detailed description of methodology This is a parallel-group randomized controlled trial, blinded to the 17β-estradiol (n=10) or placebo (n=10) supplement administered every day for 10 days. Twelve healthy young men (age: 18-25yrs; BMI: 22-33 kg/m2) will be recruited to participate in this study. During phone or e-mail conversations we will explain the purpose and experimental design of the study and address all questions the participants might have (see telephone and email scripts). Participants will visit the laboratory for a screening to assess whether they are eligible to participate in this study. During the screening we will first explain the experimental design and obtain written informed consent. A medical questionnaire will be completed by the participants to assess their general health and use of medication. Body height and mass will be measured as baseline characteristics of the participants. Participants will be requested to fill out a 3-d dietary record to assess habitual energy and protein intake. Participants will be randomly assigned to the 17β-estradiol (n=10) or placebo (n=10) supplementation group. Randomization will be performed using a computerized list randomizer (https://www.random.org/lists/), and participants will be sequentially allocated to a condition according to the randomized list. The experimental trial is composed of 10 days of 17β-estradiol (Estrace, Acerus Pharmaceuticals Corporation, Mississauga, ON, Canada or placebo (400 mg/day Polycose, Abbott Laboratories, St. Laurent, QC, Canada) supplementation, including 3 days of pre-immobilization, and 7 days of single leg immobilization. Three days prior to immobilization (t=-3 d) a blood sample will be obtained and muscle strength will be assessed before daily 17β-estradiol or placebo supplementation will be initiated. Participants will consume 1mg/day for 3-days and 3mg/day for 7-days of Estrace or 400 mg/day of Polycose for 7-days. The estrogen and placebo bottles are coded to ensure complete blinding to both researchers and participants. Additional blood samples will be obtained to assess the compliance of the participants to the supplementation. In addition, at t=-3 d a saliva sample will be obtained before ingesting 150 mL of deuterium-labeled water (D2O). Daily saliva sampling will be continued until the end of the experimental trial to assess precursor pool enrichments. Dietary intake will be controlled for 10-days (including 3 d prior to immobilization and 7 d of immobilization) providing an energy balanced diet containing 1 weight per day equally distributed over breakfast, lunch, and dinner (15). Participants will be instructed to refrain from vigorous-intensity physical activity (running, fast cycling, competitive sports, carrying heavy loads, etc.) and refrain from alcohol consumption for 3 d prior to and during the 7-day single leg immobilization. Daily activity will be monitored with a SenseWear Armband, which subjects will be required to wear from t=-3 d until the end of the experimental trial.

Participants will have one leg immobilized by means of knee bracing (http://www.breg.com/products/knee-bracing/post-op) thus the contralateral limb will act as an internal control. The leg to be immobilized will be chosen in a random counterbalanced manner to result in equal numbers of participants having their weaker or stronger legs being immobilized. The brace (http://www.breg.com/products/knee-bracing/post-op) will be worn in a fixed flexion position at 140° (i.e., 40° from full extension) with a plastic band that is removed to check for pressure points daily and resealed with a custom-modified plastic strap that is melted to seal the strap, as we have done previously19,20. The reason for this is that the brace cannot be removed without breaking the plastic seal, but could be broken in the case of an emergency and the brace removed entirely, if required. Using this model of disuse we have found the immobilizing brace to be well tolerated, not restrictive, and importantly it does not occlude for popliteal and/or femoral artery blood flow, and we have had no cases of edema or venous thrombosis in previous studies. Participants will also be provided with elastic support bandages to lessen the risk of deep vein thrombosis.

On t=0 d, a blood sample, saliva sample and muscle biopsy will be collected for the assessment of muscle protein synthesis rates. Muscle strength and volume will be assessed using a Biodex and ultrasonography respectively. A knee brace will be placed to start the 7-day single leg immobilization phase. The choice of leg for immobilization will be randomized and balanced for dominance according to maximal isometric strength. At the end of the immobilization phase (t=7 d), a blood sample will be obtained, muscle biopsies will be collected from both the immobilized and non-immobilized leg, and muscle volume and strength will be assessed. After strength is assessed in both legs, a further muscle biopsy will be taken to assess the effect of 17β-estradiol on muscle response to a single bout of exercise (Biodex) in both the non-immobilized and immobilized leg 3-hrs after the exercise bout.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy, non-smoking as assessed by questionnaire
2. Willing and able to provide informed consent
3. BMI between 22 and 29 kg/m2

Exclusion Criteria:

1. Any concurrent medical, orthopedic, or psychiatric condition that, in the opinion of the Investigators, would compromise the ability to comply with the study requirements
2. Significant orthopedic, cardiovascular, pulmonary, renal, liver, infectious disease, immune disorder, or metabolic/endocrine disorders or other disease that would preclude oral 17β-estradiol supplementation
3. Current illnesses which could interfere with the study (e.g. prolonged severe diarrhea, regurgitation, difficulty swallowing)
4. Excessive alcohol consumption (>21 units/week)
5. History of bleeding diathesis, platelet or coagulation disorders, or antiplatelet/anticoagulation therapy
6. Personal or family history of clotting disorder or deep vein thrombosis
7. Concomitant use of corticosteroids, testosterone replacement therapy (ingestion, injection, or transdermal), or any anabolic steroid

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-05 (Estimated); Primary Completion 2018-05 (Estimated); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Muscle protein synthesis and breakdown rates | Prior to immobilization (-3-0 d) and over the 7 days of immobilization (0-7 d).
  Myofibrillar protein will be extracted from the muscle biopsies. Myofibrillar protein-bound 2H-alanine enrichments will be determined by gas chromatography-combustion-isotope ratio mass spectrometry (GC-C-IRMS) by Metabolic Solutions, Nashua, NH as described previously (16). The saliva and plasma samples will be analyzed for 2H enrichments by cavity ring-down spectroscopy by Metabolic Solutions. Fractional synthetic rates of muscle protein synthesis will be calculated by dividing the increment in muscle protein-bound enrichment between two muscle biopsies over time by the average enrichment in total body water/plasma.

SECONDARY OUTCOMES:
Muscle size | At t=0 and after 7 days of immobilization.
  Ultrasound will be performed on both legs to assess leg muscle volume and mass.
Muscle strength | At t=0 and after 7 days of immobilization.
  Muscle strength will be assessed using Biodex.

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Phillips, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster Univeristy, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No